CLINICAL TRIAL: NCT01696357
Title: Developing an Automated Symptom Monitoring Device for Adolescents With Asthma
Brief Title: Automated Device for Asthma Monitoring
Acronym: ADAM
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hyekyun Rhee, Associate Professor, University of Rochester
Other Study IDs: 5R01NR011169 (NIH)
Record Dates: First submitted 2012-09-18; First posted 2012-10-01 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: Asthma; Adolescents; Self-monitoring; Quality of life; Biomedical device; Symptom monitoring; Self-management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adolescents with asthma: Ages 13-17 with an asthma diagnosis-both symptomatic and non-symptomatic- and with currently prescribed asthma medication.
  Interventions: Device: Automated Device for Asthma Monitoring (ADAM)
- Adolescents without asthma: Ages 13-17 without an asthma diagnosis and without any other respiratory condition that presents with asthma-like symptoms.
  Interventions: Device: Automated Device for Asthma Monitoring (ADAM)

INTERVENTIONS:
Device: Automated Device for Asthma Monitoring (ADAM) — Both groups of adolescents (asthma/non-asthma)wore a prototype ADAM device for 7 days as they went about their usual daily activities. At night, the device continued to monitor symptoms as it was placed in close proximity to the adolescent's head during sleep. The asthma group answered survey questions about the status of their symptoms and their usage of asthma medication every morning and every evening- entering their answers directly onto the monitoring device.

SUMMARY:
This study will examine an innovative strategy to monitor asthma symptoms by using existing technology to develop a non-invasive device for monitoring asthma symptoms in adolescents. Using an iPod as a platform, and current sound data analysis techniques, a prototype device will be developed that will directly monitor the chosen parameters of asthma symptoms, including wheezing, coughing and activity levels. This small non-invasive device will be continuously carried by or placed in close proximity to the adolescent on a daily basis. It is hypothesized that such a device would be acceptable to adolescents and would lend accuracy and objectivity to symptom assessment; something that existing monitoring strategies have yet to achieve. It will also stimulate the adolescents' partnership in asthma self-monitoring and ultimately lead to effective asthma management.

DETAILED DESCRIPTION:
Prior research has generated compelling evidence that programs promoting self-management can reduce morbidity and improve asthma outcomes in children. Successful asthma management strategies require patients' active commitment to engage in care processes by establishing self-monitoring routines. Adequate self-monitoring of asthma symptoms is considered to be the cornerstone of appropriate asthma management leading to fewer cases of asthma exacerbation and acute care visits as well as better functional outcomes and higher quality of life in children and adolescents. Symptom monitoring informs patient decisions to initiate necessary self-management behaviors (e.g., adjust medication, alter activity level, alter the surrounding environment or seek medical assistance) as well as the providers' decisions related to an appropriate treatment course such as step up, no change or step down therapy. Thus, current guidelines by National Heart, Lung, and Blood Institute (NHLBI) Expert Panel Review 3 (EPR3) highlight the importance of ongoing symptom monitoring.

Studies of children have raised concerns about adequacy and effectiveness of current methods of asthma self-monitoring including symptom-based and peak expiratory flow (PEF) monitoring. Symptom-based monitoring relies on the individual's symptom perception which is subjective and influenced by a variety of factors such as the patient's emotional status, social influences (e.g, family, peers) and previous experiences with symptoms. Thus, the accuracy and objectivity of this monitoring method is uncertain. As an objective approach, PEF monitoring has been encouraged, yet the efficacy of this method has also been a subject of ongoing debate in the literature. Poor adherence and inadequate technique further diminish the clinical usefulness of PEF monitoring. Thus, the uncertainty of current monitoring strategies underscores the imperative of an alternative symptom monitoring strategy that addresses the issues of accuracy and objectivity of symptom assessment.

Adolescence is an important period for consolidating and establishing self-management of and adjustment to chronic health conditions. Yet an array of developmental challenges including the desire for normalcy and peer approval, feelings of invulnerability and emerging independence undermine adolescents' motivation and behaviors to engage in self-management and present particular difficulties in achieving optimal asthma control in adolescents with asthma. Parents become less able to manage asthma as children reach adolescence and many researchers and clinicians have reported similar difficulties in managing asthma in adolescents primarily due to inadequate adherence and counterproductive behaviors. Thus, clinicians face serious challenges in providing optimal management for adolescents with asthma primarily due to difficulties in soliciting patients' active partnership in asthma management with sustainable and reliable symptom monitoring routines. Accurate symptom monitoring by patients is the most fundamental antecedent to effective asthma management, yet existing monitoring strategies have not been conducive to adolescents' cooperation or yielded accurate or clinically useful information. Having recognized these limitations, this study will examine an innovative strategy to monitor asthma symptoms that stimulates adolescents' partnership and ultimately leads to effective asthma management.

The device will directly monitor the chosen parameters of asthma symptoms, including wheezing, coughing and activity levels. A mobile phone will be employed as a platform for processing, analyzing and storing data transmitted from a microphone and a wireless accelerometer. This new approach is developmentally appropriate, given adolescents' affinity for technology and its capacity to address adolescents' need for maintaining normalcy while allowing continuous asthma monitoring during real-life situations. The device involves biomedical engineering techniques enabling automatic sound and activity recording, analysis, feedback, and storage function. A mobile phone will be employed as a platform for processing, analyzing and storing data transmitted from a microphone and a wireless accelerometer. This technology will automate daily symptom monitoring with minimal intrusiveness and maximum accuracy, thereby reducing the risk of inappropriate treatment and ameliorating asthma-related disability. Due to its foreseen safety, noninvasiveness, objectivity, convenience, user-friendliness, and cost containment, the approach can greatly enhance asthma management by adolescents and health care providers. This device has the potential to bring about patient behavior changes such as avoiding triggers and adjusting medications as the device will provide the opportunity for in-time review of symptoms.

ELIGIBILITY:
Inclusion Criteria: Asthma Group

* Age 13 through 17 years,
* Asthma diagnosis from a care provider,
* Prescribed asthma controller medication

Inclusion Criteria: Comparison(Non-asthma)Group

* Age 13 through 17 years,

Exclusion Criteria: Asthma Group

* Other health conditions (e.g., heart disease, cystic fibrosis) producing asthma-like symptoms,
* Known cognitive, psychological and behavior problems (based on self-report and/or clinician report) that present challenges in following study procedures
* Ability to understand spoken and written English.

Exclusion Criteria: Comparison(Non-asthma)Group

* Other health conditions (e.g., heart disease, cystic fibrosis) producing asthma-like symptoms,
* Known cognitive, psychological and behavior problems (based on self-report and/or clinician report) that present challenges in following study procedures
* Ability to understand spoken and written English.
* Asthma diagnosis from a care provider,

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents between the ages of 13-17 who received care at Strong Memorial Hospital, Rochester NY.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyekyun Rhee, PhD, RN, PNP, Principal Investigator — University of Rochester School of Nursing; Mark Bocko, PhD, Principal Investigator — University of Rochester Electrical Engineering
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Rhee H, Miner S, Sterling M, Halterman JS, Fairbanks E. The development of an automated device for asthma monitoring for adolescents: methodologic approach and user acceptability. JMIR Mhealth Uhealth. 2014 Jun 19;2(2):e27. doi: 10.2196/mhealth.3118. PMID 25100184
- [Result] Rhee H, Fairbanks E, Butz A. Symptoms, feelings, activities and medication use in adolescents with uncontrolled asthma: lessons learned from asthma diaries. J Pediatr Nurs. 2014 Jan-Feb;29(1):39-46. doi: 10.1016/j.pedn.2013.04.009. Epub 2013 May 15. PMID 23685266
- [Result] Sterling M, Rhee H, Bocko M. Automated Cough Assessment on a Mobile Platform. J Med Eng. 2014;2014:951621. doi: 10.1155/2014/951621. PMID 25506590
- [Derived] Rhee H, Belyea M, Mammen J. Visual analogue scale (VAS) as a monitoring tool for daily changes in asthma symptoms in adolescents: a prospective study. Allergy Asthma Clin Immunol. 2017 Apr 28;13:24. doi: 10.1186/s13223-017-0196-7. eCollection 2017. PMID 28465694

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adolescents With Asthma | Adolescents Without Asthma
Started | 42 | 42
Completed | 40 | 41
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents With Asthma | Adolescents Without Asthma | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.5) | 14.8 (1.3) | 15.0 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Coughs Per Hour
Description: The device is supposed to detect and count the number of coughs per 24 hours and register the numbers into the device.
Time Frame: 7 days
Population: One subject in the non-asthma group failed to return the device after the 7-trial. Data from 22 participants (3 from the asthma group, 19 from non-asthma group) were not included in the analysis as no data were recorded (due to a mechanical issue) or data were too extreme (due to cough algorithm failure).
Measure: Mean (Standard Deviation); unit: average number of coughs per hour
Arm/Group | Adolescents With Asthma | Adolescents Without Asthma
Number analyzed (Participants) | 39 | 22
average number of coughs per hour | 57.64 (111.41) | .63 (.76)

ADVERSE EVENTS:
Arm/Group | Adolescents With Asthma | Adolescents Without Asthma
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No